CLINICAL TRIAL: NCT03068169
Title: Biomedical Shirt-based ECG Monitoring in Relevant Clinical Situations
Brief Title: Biomedical Shirt-based ECG Monitoring
Acronym: ECG-shirt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marcin Grabowski, Clinical Professor, Medical University of Warsaw
Other Study IDs: ECG-shirt study
Record Dates: First submitted 2017-02-10; First posted 2017-03-01 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: ECG Monitoring
Keywords: remote ECG; atrial fibrillation; cardiac rehabilitation; cardiac resynchronization therapy; supraventricular tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular diseases (CVD) are associated with high healthcare costs, as well as are a leading cause of mortality and hospitalizations. The main challenge for today's researchers is to develop new technologies, which may help to improve diagnosis of CVD, thereby reducing healthcare costs and quality of patients' lives. Non-invasive wearable electronics offer new capabilities for the diagnosis and management of patients with CVD. Several reports with wearable electronics have been published, in which achieved very positive results with high accuracy. Aim of our study is to show utility of biomedical shirt-based ECG monitoring of patients with CVD in different clinical situations using Nuubo® ECG (nECG) system.

DETAILED DESCRIPTION:
The study is an investigator-initiated, multicentre, prospective observational trial. The study will be carried out in 2 tertiary university hospitals on cardiology wards (adult and pediatric). The study will consist of four independent groups of patients whose ECG will be monitored using the biomedical shirt. The study groups will be as follows: patients after pulmonary veins isolation (PVI), cardiac resynchronization therapy (CRT) recipients, patients during cardiac rehabilitation after myocardial infarction, and pediatric patients with supraventricular tachycardia (SVT) before electrophysiology study (EPS). Approval for all study groups was obtained from institutional review board.

ECG platform The system consists of biomedical shirt, electronic device and ECG software. The biomedical shirt captures the electrocardiographic signal via the textile electrodes integrated into the garment. The biomedical shirt enable non-invasive reception of a medical-quality ECG signal through adherence of textile electrodes to the skin. The biomedical shirt-ECG monitoring is based on BlendFix® sensor electrode technology that is capable of being used in real-time and for continuous recording. To the shirt is attached the electronic device that transmits the ECG signal (as well as other signals including accelerometer and GPS) via bluetooth to a computer and stores the information in memory cards. The software allows the visualisation and analysis of data such as ECG, heart rate, activity index and relative position of the body captured by the electronic device. The platform is a medical device certified in the European Union that has been tested in patients who underwent an exercise echocardiography test.

ELIGIBILITY:
Patients after PVI

Inclusion Criteria:

* PVI in a patient with paroxysmal AF
* 18 - 70 years old
* Signed written informed consent Exclusion criteria
* BMI ≥35 kg/m2
* Chronic inflammatory disease, severe chronic kidney disease,
* Active cancer, and a period of 5 years from the end of treatment
* Use of antiarrhythmic agents after PVI
* Persistent AF
* Previous PVI
* The size of the chest that prevents wearing biomedical shirt
* Contraindications to wear biomedical shirt (structural disease of the chest, skin diseases, allergy for materials used in ECG shirts)

CRT recipients

Inclusion criteria:

* > 18 years old
* Meeting the current European Society of Cardiology Guidelines indications for CRT implantation (including upgrades)
* Signed written informed consent Exclusion criteria
* Chest size which make impossible to wear nECG shirt
* Contraindications to wear biomedical shirt (structural disease of the chest, skin diseases, allergy for materials used in ECG shirts)

Patients during cardiac rehabilitation after myocardial infarction

Inclusion criteria:

* Patients within 3 months after myocardial infarction, after completed early post-infarction ambulatory cardiac rehabilitation
* Signed written informed consent
* 18 - 80 years old

Exclusion criteria:

* Dysfunction of the lower limbs or other walking impairments,
* Age below 18 or over 80 years old.
* Unstable angina pectoris.
* Life-threatening arrhythmias.
* Decompensated congestive heart failure.
* Left ventricular ejection fraction <35%.
* Dissecting aneurysm of the aorta.
* Acute myocardial infarction.
* Vein thrombophlebitis.
* Pulmonary or peripheral embolism.
* Uncontrolled hypertension.
* Active inflammation.
* Other contraindication to physical activity.
* The state after the pacemaker or implantable cardioverter-defibrillator implantation (contraindication to bioelectrical impedance measurement).
* Persistent AF
* Previous PVI

Pediatric patients with SVT

Inclusion criteria:

* 5-18 years old
* Patients with diagnosed SVT qualified to EPS
* Signed written informed consent

Exclusion criteria:

* BMI ≥35 kg/m2
* Chronic inflammatory disease, severe chronic kidney disease,
* Active cancer, and a period of 5 years from the end of treatment
* The size of the chest that prevents wearing biomedical shirt
* Contraindications to wear biomedical shirt (structural disease of the chest, skin diseases, allergy for materials used in ECG shirts)

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be consisted of four independent patient groups: 30 patients with paroxysmal AF treated with PVI; 30 patients scheduled for CRT implantation; 120 patients after early post-infarction ambulatory cardiac rehabilitation; 40 patients, between 5 to 18 years old, with diagnosed SVT and who are qualified for electrophysiological study (EPS).
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between early recurrences of atrial tachyarrhythmias (ERAT) during blanking period on long-term effectiveness of pulmonary veins isolation (PVI) using nECG shirt. | 13 months
  Assessment of the rationale for the use of blanking period and to determine whether the early recurrences of atrial tachyarrhythmias (ERAT) burden influences on long-term effectiveness of pulmonary veins isolation (PVI) using nECG shirt. The study might demonstrate which patients with ERAT remain at risk of long-term recurrence of atrial fibrillation (AF).
Assessment of the usefulness of nECG shirt in detection of fusion and pseudo-fusion beats in cardiac resynchronization therapy (CRT) recipients. | 7 months
Assessment of the impact of the use of a pedometer combined with nECG shirt on the level of daily physical activity and its intensity. | 12 month
Creation of an algorithm based on nECG monitoring using wearable shirt to differentiate atrioventricular reentry tachycardia (AVRT) with atrioventricular nodal reentry tachycardia (AVNRT) in pediatric patients suffering from supraventricular tachycardia. | 1 month

SECONDARY OUTCOMES:
Assessment of the influence of CRT implantation on amount of physical activity measured by nECG shirt. | 7 month

CONTACTS AND LOCATIONS:
Overall Officials: Renata Główczyńska, PhD, Principal Investigator — 1st Department of Cardiology Medical University of Warsaw; Paweł Balsam, PhD, Principal Investigator — 1st Department of Cardiology Medical University of Warsaw; Piotr Lodziński, PhD, Principal Investigator — 1st Department of Cardiology Medical University of Warsaw; Marcin Grabowski, PhD, Principal Investigator — 1st Department of Cardiology Medical University of Warsaw
Locations (3):
- Poland (3):
  - Department of Pediatric Cardiology and General Pediatrics, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Department of Clinical Nursing, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Paweł Balsam, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for meta-analysis

REFERENCES:
- [Derived] Balsam P, Lodzinski P, Tyminska A, Ozieranski K, Januszkiewicz L, Glowczynska R, Wesolowska K, Peller M, Pietrzak R, Ksiazczyk T, Borodzicz S, Koltowski L, Borkowski M, Werner B, Opolski G, Grabowski M. Study design and rationale for biomedical shirt-based electrocardiography monitoring in relevant clinical situations: ECG-shirt study. Cardiol J. 2018;25(1):52-59. doi: 10.5603/CJ.a2017.0102. Epub 2017 Aug 25. PMID 28840587